CLINICAL TRIAL: NCT01263509
Title: A Long-term, Open-label Extension Study to Investigate the Long-term Safety of SYR-322 When Used in Combination With α-glucosidase Inhibitor in Subjects With Type 2 Diabetes in Japan
Brief Title: Long-term Safety Study of Alogliptin Used in Combination With α-glucosidase Inhibitor in Participants With Type 2 Diabetes in Japan
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SYR-322/OCT-003; U1111-1118-3992 (Registry Identifier: WHO)
Record Dates: First submitted 2010-12-17; First posted 2010-12-20 (Estimated); Results first posted 2011-08-29 (Estimated); Last update posted 2012-02-03 (Estimated); Status verified 2012-02

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Diabetes Mellitus - Type 2; Diabetes Mellitus; Drug Therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — alogliptin; voglibose

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID (Experimental)
  Interventions: Drug: Alogliptin and voglibose
- Alogliptin 25 mg QD and Voglibose 0.2 mg TID (Experimental)
  Interventions: Drug: Alogliptin and voglibose

INTERVENTIONS:
Drug: Alogliptin and voglibose — Alogliptin 12.5 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  Other Names: SYR-322; Voglibose; BASEN®
  Arms: Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID
Drug: Alogliptin and voglibose — Alogliptin 25 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  Other Names: SYR-322; Voglibose; BASEN®
  Arms: Alogliptin 25 mg QD and Voglibose 0.2 mg TID

SUMMARY:
The purpose of this study was to evaluate the long-term safety and efficacy of alogliptin and an α-glucosidase inhibitor administered once daily (QD) or three times daily (TID) for 40 consecutive weeks in participants who completed a phase 2/3 α-glucosidase inhibitor add on study.

DETAILED DESCRIPTION:
Both insulin hyposecretion and insulin-resistance are considered to be involved in the development of type 2 diabetes mellitus.

Takeda is developing SYR-322 (alogliptin) for the improvement of glycemic control in patients with type 2 diabetes mellitus. Alogliptin is an inhibitor of the dipeptidyl peptidase IV (DPP-IV) enzyme. DPP-IV is thought to be primarily responsible for the degradation of 2 peptide hormones released in response to nutrient ingestion. It is expected that inhibition of DPP-IV will improve glycemic control in patients with type 2 diabetes.

"To evaluate the long-term safety and efficacy of alogliptin and an α-glucosidase inhibitor, this extension study was administered for 40 consecutive weeks (52 weeks from the start of treatment in the phase 2 dose-ranging study) to participants who completed a phase 2/3 α-glucosidase inhibitor add on study 322/CCT-003 (NCT01263483).

ELIGIBILITY:
Inclusion Criteria:

* Had completed the phase 2 dose-ranging study (i.e., the subject had completed the study visit at Week 12).

Exclusion Criteria:

* Had clinical manifestations of hepatic impairment (e.g., an aspartate aminotransferase or alanine aminotransferase value 2.5 times or more of the upper reference limit at Week 8 of treatment in the phase 2 dose-ranging study).
* Had clinical manifestations of renal impairment (e.g., a creatinine value of 2 mg/dL or more at Week 8 of treatment in the phase 2 dose-ranging study).

Ages: 33 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 179 (Actual)
Dates: Start 2007-06; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Department of Medicine, Study Director — Kawasaki Medical School

REFERENCES:
- [Derived] Seino Y, Fujita T, Hiroi S, Hirayama M, Kaku K. Alogliptin plus voglibose in Japanese patients with type 2 diabetes: a randomized, double-blind, placebo-controlled trial with an open-label, long-term extension. Curr Med Res Opin. 2011 Nov;27 Suppl 3:21-9. doi: 10.1185/03007995.2011.614936. PMID 22106975

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled at 24 investigative sites in Japan from 06 June 2007 to 02 October 2008.
Pre-assignment Details: Participants enrolled in one of 2, once-daily (QD) or three-times daily (TID) treatment groups. Analyses performed by treatment group or treatment dose in this study. All 213 participants randomized in the phase 2/3 α-glucosidase inhibitor (NCT01263483) study are included in the Full Analysis Set in this study, of which 179 randomized.
Groups:
- 12.5 mg Combination Dose Group* → 12.5 mg Combination Group: Alogliptin 12.5 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the 12.5 mg combination dosing ARM of the SYR-322/CCT-003 (NCT01263483) core phase 2/3 add on study.
- 25 mg Combination Dose Group* → 25 mg Combination Dose Group: Alogliptin 25 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the for 25 mg combination dosing ARM of the SYR-322/CCT-003 (NCT01263483) core phase 2/3 add on study.
- α-glucosidase Monotherapy Group* → 12.5 mg Combination Group: Alogliptin 12.5 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the α-glucosidase inhibitor monotherapy dosing ARM of the SYR-322/CCT-003 (NCT01263483) core phase 2/3 add on study.
- α-glucosidase Monotherapy Group*→ 25 mg Combination Group: Alogliptin 25 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
  *for participants from the α-glucosidase inhibitor monotherapy dosing ARM of the SYR-322/CCT-003 (NCT01263483) core phase 2/3 add on study.
Period: Enrolled - Long-Term Extension Study
Arm/Group | 12.5 mg Combination Dose Group* → 12.5 mg Combination Group | 25 mg Combination Dose Group* → 25 mg Combination Dose Group | α-glucosidase Monotherapy Group* → 12.5 mg Combination Group | α-glucosidase Monotherapy Group*→ 25 mg Combination Group
Started | 61 | 60 | 32 | 26
Completed | 61 | 60 | 32 | 26
Not Completed | 0 | 0 | 0 | 0
Period: Entered - Long-Term Extension Study
Arm/Group | 12.5 mg Combination Dose Group* → 12.5 mg Combination Group | 25 mg Combination Dose Group* → 25 mg Combination Dose Group | α-glucosidase Monotherapy Group* → 12.5 mg Combination Group | α-glucosidase Monotherapy Group*→ 25 mg Combination Group
Started | 61 | 60 | 32 | 26
Completed | 53 | 48 | 27 | 24
Not Completed | 8 | 12 | 5 | 2
Not completed — Adverse Event | 5 | 5 | 4 | 1
Not completed — Lack of Efficacy | 1 | 4 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0 | 0
Not completed — Participant Unavailability | 1 | 1 | 0 | 0
Not completed — Poor Glycosylated Hemoglobin Control | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID: Alogliptin 12.5 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
- Alogliptin 25 mg QD and Voglibose 0.2 mg TID: Alogliptin 25 mg, tablets, orally, once daily and voglibose 0.2 mg, tablets, orally, three times daily for up to 40 weeks.
- Total: Total of all reporting groups
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID | Total
Number analyzed (Participants) | 108 | 105 | 213
Age, Customized [Number; unit: participants]
  ≤ 64 years | 69 | 53 | 122
  ≥ 65 years | 39 | 52 | 91
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 38 | 82
  Male | 64 | 67 | 131

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events.
Description: A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug and within 30 days after receiving the last dose of study drug. A TEAE may also be a pre-treatment adverse event or a concurrent medical condition diagnosed prior to the date of first dose of study drug, which increases in intensity after the start of dosing. Adverse events data with onset occurring more than 30 days after last dose of study drug (AE start date - last dose date >30) will be listed, but not included in the summary tables below.
Time Frame: 52 Weeks.
Population: Adverse Event Profile in the Safety Analysis Set
Measure: Number; unit: participants
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 108 | 105
participants
  Serious Adverse Event | 6 | 7
  Serious Adverse Event Related to Study Drug | 0 | 1
  Other Adverse Events (Incidence ≥3%) | 85 | 73

2. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 8).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 8 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 8.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 107 | 100
percentage of Glycosylated Hemoglobin | -0.69 (0.479) | -0.79 (0.417)

3. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 12).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 12 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 99
percentage of Glycosylated Hemoglobin | -0.89 (0.589) | -0.96 (0.486)

4. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 16).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 16 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 16.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 91 | 84
percentage of Glycosylated Hemoglobin | -0.91 (0.658) | -0.96 (0.587)

5. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 20).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 20 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 20.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 90 | 83
percentage of Glycosylated Hemoglobin | -0.90 (0.745) | -0.89 (0.592)

6. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 24).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 24 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 90 | 82
percentage of Glycosylated Hemoglobin | -0.83 (0.750) | -0.88 (0.624)

7. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 28).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 28 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 28.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 88 | 82
percentage of Glycosylated Hemoglobin | -0.81 (0.704) | -0.89 (0.619)

8. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 32).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 32 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 32.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 86 | 82
percentage of Glycosylated Hemoglobin | -0.80 (0.701) | -0.85 (0.679)

9. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 36).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 36 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 36.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 84 | 78
percentage of Glycosylated Hemoglobin | -0.82 (0.717) | -0.90 (0.649)

10. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 40).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 40 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 40.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 82 | 78
percentage of Glycosylated Hemoglobin | -0.78 (0.742) | -0.92 (0.672)

11. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 44).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 44 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 44.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 53 | 51
percentage of Glycosylated Hemoglobin | -0.88 (0.721) | -0.94 (0.545)

12. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 48).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 48 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 48.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 53 | 49
percentage of Glycosylated Hemoglobin | -0.92 (0.694) | -0.94 (0.548)

13. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Week 52).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 52 and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 53 | 48
percentage of Glycosylated Hemoglobin | -0.95 (0.692) | -0.95 (0.568)

14. Secondary Outcome: Change From Baseline in Glycosylated Hemoglobin (Final Visit).
Description: The change in the value of glycosylated hemoglobin (the concentration of glucose bound to hemoglobin as a percent of the absolute maximum that can be bound) collected at week 52 or final visit and glycosylated hemoglobin collected at baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: percentage of Glycosylated Hemoglobin
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 108 | 105
percentage of Glycosylated Hemoglobin | -0.81 (0.714) | -0.89 (0.660)

15. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 8).
Description: The change between the value of fasting plasma glucose collected at week 8 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 8.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 107 | 100
mg/dL | -18.2 (22.43) | -20.4 (23.04)

16. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 12).
Description: The change between the value of fasting plasma glucose collected at week 12 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 99
mg/dL | -17.1 (22.02) | -18.8 (24.26)

17. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 16).
Description: The change between the value of fasting plasma glucose collected at week 16 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 16.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 91 | 84
mg/dL | -16.0 (23.84) | -15.3 (23.33)

18. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 20).
Description: The change between the value of fasting plasma glucose collected at week 20 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 20.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 90 | 83
mg/dL | -15.6 (23.90) | -15.0 (26.34)

19. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 24).
Description: The change between the value of fasting plasma glucose collected at week 24 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 90 | 82
mg/dL | -13.8 (23.96) | -15.6 (26.84)

20. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 28).
Description: The change between the value of fasting plasma glucose collected at week 28 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 28.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 88 | 82
mg/dL | -14.5 (22.77) | -21.9 (23.68)

21. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 32).
Description: The change between the value of fasting plasma glucose collected at week 32 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 32.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 86 | 82
mg/dL | -17.7 (20.75) | -20.1 (29.84)

22. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 36).
Description: The change between the value of fasting plasma glucose collected at week 36 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 36.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 83 | 78
mg/dL | -17.3 (22.93) | -22.6 (27.10)

23. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 40).
Description: The change between the value of fasting plasma glucose collected at week 40 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 40.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 82 | 78
mg/dL | -19.7 (22.88) | -22.8 (23.49)

24. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 44).
Description: The change between the value of fasting plasma glucose collected at week 44 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 44.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 53 | 51
mg/dL | -21.5 (19.63) | -24.4 (26.01)

25. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 48).
Description: The change between the value of fasting plasma glucose collected at week 48 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 48.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 53 | 49
mg/dL | -20.5 (21.12) | -23.1 (27.16)

26. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Week 52).
Description: The change between the value of fasting plasma glucose collected at week 52 and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 53 | 48
mg/dL | -20.7 (20.37) | -24.0 (20.98)

27. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (Final Visit).
Description: The change between the value of fasting plasma glucose collected at week 52 or final visit and fasting plasma glucose collected at baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 108 | 105
mg/dL | -17.5 (23.45) | -23.3 (26.35)

28. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 8).
Description: The change between the value of fasting C-peptide collected at week 8 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 8.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 107 | 100
ng/mL | 0.05 (0.701) | 0.11 (0.680)

29. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 12).
Description: The change between the value of fasting C-peptide collected at week 12 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 99
ng/mL | 0.10 (0.743) | 0.13 (0.603)

30. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 16).
Description: The change between the value of fasting C-peptide collected at week 16 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 16.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 91 | 84
ng/mL | 0.24 (0.761) | 0.21 (0.597)

31. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 20).
Description: The change between the value of fasting C-peptide collected at week 20 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 20.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 87 | 83
ng/mL | 0.24 (0.840) | 0.15 (0.801)

32. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 24).
Description: The change between the value of fasting C-peptide collected at week 24 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 81 | 76
ng/mL | 0.19 (0.897) | 0.14 (0.723)

33. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 28).
Description: The change between the value of fasting C-peptide collected at week 28 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 28.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 70 | 71
ng/mL | 0.18 (0.984) | 0.25 (0.788)

34. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 32).
Description: The change between the value of fasting C-peptide collected at week 32 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 32.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 58 | 63
ng/mL | 0.47 (0.895) | 0.31 (0.799)

35. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 36).
Description: The change between the value of fasting C-peptide collected at week 36 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 36.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 37 | 39
ng/mL | 0.33 (0.695) | 0.38 (0.654)

36. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 40).
Description: The change between the value of fasting C-peptide collected at week 40 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 40.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 28 | 28
ng/mL | 0.30 (0.701) | 0.37 (0.604)

37. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 44).
Description: The change between the value of fasting C-peptide collected at week 44 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 44.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 11 | 13
ng/mL | 0.08 (0.698) | 0.25 (0.477)

38. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 48).
Description: The change between the value of fasting C-peptide collected at week 48 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 48.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 4 | 4
ng/mL | 0.45 (0.058) | 0.38 (0.340)

39. Secondary Outcome: Change From Baseline in Fasting C-peptide (Week 52).
Description: The change between the value of fasting C-peptide collected at week 52 and fasting C-peptide collected at baseline.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 3 | 1
ng/mL | 0.80 (0.600) | 0.40

40. Secondary Outcome: Change From Baseline in Fasting C-peptide (Final Visit).
Description: The change between the value of fasting C-peptide collected at week 52 or final visit and fasting C-peptide collected at baseline.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 108 | 105
ng/mL | 0.31 (0.821) | 0.29 (0.879)

41. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value) (Week 12).
Description: The change between the value of blood glucose collected at week 12 and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 100
mg/dL | 41.2 (25.19) | 37.6 (32.67)

42. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value) (Week 24).
Description: The change between the value of blood glucose collected at week 24 and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 62 | 58
mg/dL | 38.0 (29.04) | 37.1 (33.84)

43. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value) (Week 52).
Description: The change between the value of blood glucose collected at week 52 and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 82 | 77
mg/dL | 39.0 (25.71) | 40.8 (29.49)

44. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (2-hr Postprandial Value) (Final Visit).
Description: The change between the value of blood glucose collected at week 52 or final visit and blood glucose collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 101
mg/dL | 39.6 (26.16) | 39.4 (29.46)

45. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)) (Week 12).
Description: as for outcome 41
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg•hr/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 105 | 98
mg•hr/dL | -73.2 (63.40) | -76.8 (58.92)

46. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)) (Week 24).
Description: as for outcome 42
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg•hr/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 62 | 58
mg•hr/dL | -69.0 (61.21) | -70.4 (68.54)

47. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)) (Week 52).
Description: as for outcome 43
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg•hr/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 81 | 76
mg•hr/dL | -83.5 (58.30) | -83.4 (53.80)

48. Secondary Outcome: Change From Baseline in Blood Glucose Measured by Meal Tolerance Testing (AUC (0-2)) (Final Visit).
Description: as for outcome 44
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: mg•hr/dL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 105 | 99
mg•hr/dL | -77.5 (61.67) | -82.2 (62.58)

49. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2)) (Week 12).
Description: The change between the value of insulin collected at week 12 and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: μU•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 99 | 92
μU•hr/mL | 3.05 (15.254) | 2.95 (15.704)

50. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2)) (Week 24).
Description: The change between the value of insulin collected at week 24 and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: μU•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 59 | 55
μU•hr/mL | 4.42 (13.445) | 2.26 (13.455)

51. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2)) (Week 52).
Description: The change between the value of insulin collected at week 52 and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: μU•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 75 | 71
μU•hr/mL | -1.28 (10.220) | 0.18 (12.425)

52. Secondary Outcome: Change From Baseline in Insulin Measured by Meal Tolerance Testing (AUC(0-2)) (Final Visit).
Description: The change between the value of insulin collected at week 52 or final visit and insulin collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: μU•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 99 | 93
μU•hr/mL | -0.61 (11.454) | 0.01 (12.567)

53. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2)) (Week 12).
Description: The change between the value of C-peptide collected at week 12 and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 98
ng•hr/mL | 0.71 (2.062) | 0.71 (2.209)

54. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2)) (Week 24).
Description: The change between the value of C-peptide collected at week 24 and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 61 | 58
ng•hr/mL | 1.38 (1.845) | 1.12 (2.238)

55. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2)) (Week 52).
Description: The change between the value of C-peptide collected at week 52 and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 4 | 3
ng•hr/mL | 0.96 (1.028) | 2.18 (3.384)

56. Secondary Outcome: Change From Baseline in C-peptide Measured by Meal Tolerance Testing (AUC(0-2)) (Final Visit).
Description: The change between the value of C-peptide collected at week 52 or final visit and C-peptide collected at baseline as measured by the meal tolerance test. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 99
ng•hr/mL | 1.05 (2.089) | 0.80 (2.354)

57. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)) (Week 12).
Description: The change between the value of glucagons collected at week 12 and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 12.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: pg•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 99
pg•hr/mL | -14.3 (42.23) | -20.0 (47.18)

58. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)) (Week 24).
Description: The change between the value of glucagons collected at week 24 and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 24.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: pg•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 62 | 58
pg•hr/mL | -4.6 (53.17) | -6.8 (36.78)

59. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)) (Week 52).
Description: The change between the value of glucagons collected at week 52 and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Week 52.
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: pg•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 82 | 76
pg•hr/mL | -12.0 (64.24) | -22.2 (49.67)

60. Secondary Outcome: Change From Baseline in Glucagon Measured by Meal Tolerance Testing (AUC (0-2)) (Final Visit).
Description: The change between the value of glucagons collected at week 52 or final visit and glucagons collected at baseline. Meal tolerance test measures blood glucose, insulin, C-peptide and glucagon through blood samples drawn before a meal and 2 hours after the start of the meal.
Time Frame: Baseline and Final Visit (up to Week 52).
Population: Values are Summary Statistics.
Measure: Mean (Standard Deviation); unit: pg•hr/mL
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Number analyzed (Participants) | 106 | 100
pg•hr/mL | -11.7 (59.01) | -20.9 (50.57)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of study drug and the last dose of study drug.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID | Alogliptin 25 mg QD and Voglibose 0.2 mg TID
Serious Adverse Events (participants affected / at risk) | 6/108 | 7/105
Other Adverse Events (participants affected / at risk) | 85/108 | 73/105
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID (N=108) | Alogliptin 25 mg QD and Voglibose 0.2 mg TID (N=105)
Pneumonia (Infections and infestations) | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Angina pectoris (Cardiac disorders) | 1 | 0
Salivary gland calculus (Gastrointestinal disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alogliptin 12.5 mg QD and Voglibose 0.2 mg TID (N=108) | Alogliptin 25 mg QD and Voglibose 0.2 mg TID (N=105)
Nasopharyngitis (Infections and infestations) | 38 | 30
Bronchitis (Infections and infestations) | 6 | 3
Cystitis (Infections and infestations) | 4 | 2
Pharyngitis (Infections and infestations) | 1 | 4
Seasonal allergy (Immune system disorders) | 6 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 12 | 5
Diarrhoea (Gastrointestinal disorders) | 5 | 3
Gastritis (Gastrointestinal disorders) | 1 | 4
Abdominal distension (Gastrointestinal disorders) | 4 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 4 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 4 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 5
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 5
Gamma-glutamyltransferase increased (Investigations) | 4 | 0
Contusion (Injury, poisoning and procedural complications) | 5 | 3
Fall (Injury, poisoning and procedural complications) | 4 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The clinical trial contract states that information should never be disclosed without prior consent of the sponsor, although it does not specify the number of days during which disclosure of information is limited.